CLINICAL TRIAL: NCT03768882
Title: Comparison of the Efficacy of Intravenous Dexketoprofen and Paracetamol in the Treatment of Pain in Patients Presenting to the Emergency Department With Sore Throat: A Double-Blinded, Randomized, Controlled Trial
Brief Title: Comparison of the Efficacy of Intravenous Dexketoprofen and Paracetamol in the Treatment of Sore Throat
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Üzeyir Çimen, Research Assistant, Pamukkale University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018TPF012
Record Dates: First submitted 2018-11-21; First posted 2018-12-07 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Sore Throat
Keywords: paracetamol,dexketoprofen,emergency department,sore throat
MeSH Terms: conditions — Pharyngitis | interventions — Acetaminophen; dexketoprofen trometamol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paracetamol (Experimental): Experimental: Paracetamol 1000 mg of paracetamol (parol 10mg/ml solution Mefar,Turkey ) intravenous (IV) was given 102 patients
  Interventions: Drug: paracetamol
- dexketoprofen (Experimental): Dexketoprofen Second group: dexketoprofen 50 MG (Arveles ampoule -İE Ulagay-Menarini,Turkey) intravenous (IV) was given 98 patients
  Interventions: Drug: Dexketoprofen

INTERVENTIONS:
Drug: paracetamol — 1000 mg of paracetamol (parol 10mg/ml Mefar, Turkey) intravenous (IV) was given 102 patients
  Other Names: Perfalgan; Paracerol
  Arms: Paracetamol
Drug: Dexketoprofen — Second group: dexketoprofen 50 MG (Arveles ampoule -İE Ulagay -Menarini,Turkey) intravenous (IV) was given 98 patients
  Other Names: ASEKET; DARKIN; DEXALGIN; DESTIYO; DEXCORIL
  Arms: dexketoprofen

SUMMARY:
Currently, paracetamol and nonsteroidal antiinflammatory drugs are widely used by emergency physicians in Turkey for the treatment of sore throat. The objective of the study is compare the efficacy of intravenous dexketoprofen and paracetamol in the treatment of the pain in patients presenting to the emergency department with sore throat

DETAILED DESCRIPTION:
This is the randomized double blinded clinical trial to compare the efficacy of these two drugs in this clinical setting. A randomized clinical trial was conducted in the Emergency Department (ED) of Pamukkale University Medical Faculty Hospital Study personnel (emergency physicians and emergency service nurses) were trained before the study.

When intravenous drugs (Paracetamol, Dexketoprofen) was being recommended, an eligibility checklist was completed by the attending physician. Sore throat pain intensity scale was used to measure the severity of sore throat. According to the throat pain scale, patients with moderate-severe pain, at least 1 upper respiratory tract infection (URTI) symptom according URTI questionare, with objective findings of pharyngeal inflammation (Tonsillopharyngitis evaluation score ≥5), 60 mm or more according to the sore throat sensitivity scale (STSS), 50 mm and above according to difficulty swallowing scale (DSS), 33 mm and above according to the swollen throat scale (SwoTS) were included in the study and evaluated according to these scales.

First Group: 1000 mg of paracetamol ( parol 10mg/ml solution Mefar, Turkey) intravenous (IV) was given 100 patients, Second Group:

dexketoprofen 50 mg ( arveles ampoule -IE Ulagay-Menarini, Turkey) intravenous (IV) was given 100 patients which determined to be applied as a group.

Drug packs prepared in 150 ml serum physiology were numbered by an independent nurse, who not involved in the study Randomization was achieved by using computer software to generate random numbers. During the intervention, participants were monitored by an oxygen saturation (SpO2) monitor, an automatic sphygmomanometer (blood pressure), and a rhythm monitor (heart rate and rhythms).

Patients in both groups received two types of medication in a similarmanner, thus ensuring double blind.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sore throat less than three days
* Patients with at least one of the following:
* According to the throat pain scale, patients with moderate-severe pain,
* At least 1 upper respiratory tract infection (URTI) symptom according URTI questionare,
* Objective findings of pharyngeal inflammation (Tonsillopharyngitis evaluation score ≥5),
* 60 mm or more according to the sore throat sensitivity scale (STSS),
* 50 mm and above according to difficulty swallowing scale (DSS),
* 33 mm and above according to the swollen throat scale (SwoTS)

Exclusion Criteria:

* Patients use analgesic last 12 hours
* Patients with severe liver, kidney,pulmonary and cardiac heart failure
* To be Pregnancy and breast-feeding Patients of childbearing age who are not using a birth control method
* Patients with an allergy trait (paracetamol and dexketoprofen) Illiterates
* Patients with vision problems
* Patients use antibiotics last 24 hours
* Patients use kinolons last 7 days
* Patienst use lozange,throat spray or menthol containing products last 4 hours
* Hemodynamically unstable patients,Patients with renal transplantation
* Patients with glucose 6 phosphate dehydrogenase (G6PD) deficiency
* Patients with non-controlled hypertension
* Patients with a history of cerebrovascular disease
* Patients with Wolff-Parkinson-White syndrome or accompanying arrhythmias associated with conductive stimulus delivery in the heart

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Decreament of the pain | Baseline and 120 minutes
  Comparison of the change of sore thorat pain VAS (visual analog scale) and Sore throat relief scale score between the two groups. - (First group Paracetamol and Second Dexketoprofen)

SECONDARY OUTCOMES:
Symptom frequency | Baseline and 120 minutes
  Detection of upper respiratory tract infections symptoms frequency by using upper respiratory tract infections questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Uzeyir Cimen, MD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No